CLINICAL TRIAL: NCT04046172
Title: Treatment of Periodontal Disease in Systemic Lupus Erytematosus: A Pilot Randomized Controlled Clinical Trial
Brief Title: Treatment of Periodontal Disease in Systemic Lupus Erythematosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123436
Record Dates: First submitted 2019-07-15; First posted 2019-08-06 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Systemic Lupus Erythematosus; Periodontitis
Keywords: Periodontitis; SLE; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Periodontitis | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Intervention Model Description: Total 200 Participants for part 1 (baseline). Randomization (Part 2) Control Test group (n=15) control group (n=15)
Who Masked: Outcomes Assessor
Masking Description: It is a single-blinded study in which cardio-vascular technician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): intensive periodontal treatment (IPT)
  Interventions: Procedure: supra/sub gingival root surface debridement
- control group (Sham Comparator): Control periodontal treatment (CPT)
  Interventions: Procedure: supra-gingival scaling and polishing

INTERVENTIONS:
Procedure: supra/sub gingival root surface debridement — The test group will undergo Intensive periodontal treatment (IPT)
  Other Names: IPT
  Arms: test group
Procedure: supra-gingival scaling and polishing — Control group will receive the Control periodontal treatment (CPT).
  Other Names: CPT
  Arms: control group

SUMMARY:
The primary objective of this study is to:

Part 1 - Baseline Comparisons

The primary objective of Part 1 is to:

Investigate the association between SLE and a measures of vascular health (brachial artery flow-mediated dilatyation) in patients with Systemic Lupus Erythematosus (SLE) and a healthy periodontium compared to patients with SLE and Periodontitis (PD)

Part 2 - Pilot Randomized Clinical Trial To assess the effect of Periodontal Treatment (PT) on the endothelial function in a population of patients suffering from SLE and PD.

Secondary Secondary objectives include:

Part 1 - Baseline Comparisons

The secondary objectives of Part 1 are to investigate the association of:

* Inflammatory biomarkers in saliva and blood and periodontal status in patients with SLE and PD and those with SLE and a healthy periodontium
* The oral microbiome using plaque analysis and periodontal status in patients with SLE and PD and those with SLE and a healthy periodontium Part ParPa Part 2 - Pilot Randomized Controlled Trial Evaluate the effect of PT on biomarkers of SLE disease severity/progression in a population of patients suffering from SLE and PD.

Evaluate the effect of PT on the B cell panel in a population of patients suffering from SLE and PD.

Evaluate effect of PT on the systemic inflammatory and oxidative profile of a population of patients suffering from SLE and PD.

Evaluate effect of PT on skin lesions in a population of patients suffering from SLE and PD.

DETAILED DESCRIPTION:
The primary endpoints of this study are in two parts. One part is to quantify the vascular health in response to PD as a static point prior to active therapy compared to participants with SLE and healthy perdiodontium . The second part is to quantify and compare the clinical and systemic outcomes of cases with SLE and PD following periodontalal treamtment.

Part 1 Comparative analyses between cases (SLE with PD) and controls (SLE without PD) will be performed using ANOVA analysis. Primary outcome will be the difference in flow -mediated dilatation between groups. Multivariate analysis will be performed to adjust for a number of covariates including: age, gender, body mass index, ethnicity and supragingival plaque levels.

All secondary endpoints will be analysed with ANOVA. Pre-specified analyses of secondary outcomes will include descriptive analyses and differences.

Part 2 Primary clinical periodontal outcome will be the difference in mean flow mediated (peri-implant) at 6 months between study groups and analysed by analysis of co-variance model. Age, gender, body mass index, smoking status, ethnicity and dental plaque levels will be included as additional covariates. Pair-wise comparison and between groups differences will be calculated using Tukey HSD corrections. If the normality assumption does not seem reasonable even after transformation of original values, equivalent nonparametric methods will be used.

Primary systemic inflammatory outcome will be

Changes in FMD (primary outcome), circulating inflammatory, vascular and oxidative biomarkers (secondary outcomes) will be analysed with analysis of variance for repeated measures using a conservative F-test (Greenhouse-Geisser correction). If a treatment by time interaction will be found, pair-wise comparisons will be performed (Bonferroni-Holm adjustment). Side effects and safety data will be summarized using standard descriptive statistics. Significance will be set to be at p < 0.05.

Experimental Design

Participants will be approached by the members of healthcare research team explaining the possibilities to be included in the project. There will be limit in time (24 Hours) to decide whether participate, subject to the recruitment completion.. A sufficient number of participants meeting the necessary inclusion/exclusion criteria will be accepted for the study in order to recruit 30 patients suffering from SLE and PD. Participants who consent to this study will undergo a baseline visit (Sample size 200) in which they will have a comprehensive full mouth periodontal probing depths assessment. In addition, full mouth plaque and gingival bleeding scores will also be calculated. A series of parameters will be recorded (including age, gender, ethnicity, and body mass index). Saliva samples (1 ml) and Blood samples (32 ml) will also be collected for analysis of peripheral blood inflammatory and oxidative biomarkers. Blood cell counts, C-reactive protein, complement levels, dsDNA autoantibodies, kidney and liver function tests will also be performed. The vascular function will be assessed by means of an ultrasound scan. After randomization (selected 30 patients) to either Test or Control Group, the test group will undergo periodontal treatment in 2 sessions within a week from each other. Radiographic examination Orthopentomogram (OPG) will be taken at the second visit of patient's visit only. Optical coherence tomography will be done on the patients in vist (2,4 and 6). At 2 months both groups will be reassessed, and the same information and samples taken at baseline will be collected. The test group will undergo additional periodontal treatment visit (3) of Intensive periodontal treatment/IPT) within 3 weeks from the 2 months visit. After this visit the Control group will receive the same periodontal treatment (Control periodontal treatment/CPT). At 6 months both groups will be seen for the final study assessment. If at any of the study assessment (2 months and 6 months) participants in the control group show signs of progression of PD they will be treated separately and exited from the trial. After 6 months all the participants will have treatment irrespective of groups, if they require treatment it will provided

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female Subject must be 18 years of age or over.
2. Patients with 4 or more criteria for juvenile systemic lupus erythematosus (JSLE) or SLE according to the American College of Rheumatology (ACR) 1997 criteria or SLICC 2012 criteria or biopsy proven lupus nephritis with one additional supportive test on at least two occasions (positive Anti-nuclear antibodies (ANA), anti-dsDNA antibodies or anti-Sm antibodies).
3. Presence of moderate to severe periodontitis (at least 30 pockets with Probing depth equal or greater than 5mm).
4. Subject must have voluntarily signed the informed consent.

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. Having fewer than 15 teeth.
3. Subject knowingly has HIV or Hepatitis.
4. Subject is not capable to give informed consent.
5. Presence of concomitant rheumatoid arthritis, Sjogren syndrome, diabetes mellitus.
6. Smoking.
7. Subject on anticoagulants.
8. Subjects on chronic antibiotic therapy or who require antibiotic coverage for periodontal procedures.
9. Subjects who received periodontal treatment within 6 months from the baseline

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
To measure the effect of periodontal treatment on SLE patients | 2 years
  Endothelial function/dysfunction (vessel wall elasticity) will be observed in the population of SLE patients (30) who will undergo periodontal treatment (before and after) by using Flow mediated dilatation (FMD) which is an ultra-sound scan of brachial artery in visit 2, 4 and 6).

SECONDARY OUTCOMES:
To measure the effect of PT on biomarkers of SLE disease severity/progression in a population of patients suffering from SLE and PD. | 2 years
  30 Patients will be recruited and will run a blood test in visit 2, 4 and 6 to observe the CRP (C-reactive Protein) that is an inflammatory marker before and after Periodontal treatment in patients with SLE.
To measure the effect of Periodontal Treatment on the B-cell panel in a population of patients suffering from SLE and PD. | 2 Years
  Since B-cells (lymphocytes) are already unnaturally high in SLE patients we want to see if Periodontal Treatment decreases the total cell load/population by Flow cytometry with the blood samples taken form the (30) SLE patients in visit 2, 4 and 6.
To measure the effect of Periodontal Treatment on the systemic inflammatory and oxidative profile of a population of patients suffering from SLE and PD. | 2 years
  Because SLE and Periodontal diseases are both chronic inflammatory diseases Nitrous oxide production is raised in both diseases leading to self inflicted tissue damage. Blood will be drawn form the (30) patients with SLE and will run a D-ROM test on the blood samples taken in visit 2, 4 and 6 to observe the oxidative profile of the patients with SLE before and after periodontal treatment.
To measure the effect of Periodontal Treatment on skin lesions in a population of patients suffering from SLE and PD. | 2 years
  30 SLE patients will undergo OCT (Optical coherence tomography) investigation. SLE patients might have skin lesion as an immune destructive response by the cells. OCT will observe the skin lesions caused by the disease (SLE) in visit 2, 4 and 6 (before and after periodontal treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco D'Aiuto, PhD, Study Chair — Unit of Periodontology Eastman Dental Institute,UCL.; Coziana Ciurtin, PhD, Principal Investigator — Department of Rheumatology, UCLH.; Marco Orlandi, PhD, Study Chair — Unit of Periodontology Eastman Dental Institute,UCL.; Jacopo Buti, PhD, Study Chair — Unit of Periodontology Eastman Dental Institute,UCL.
Locations (1):
- Eastman clinical investigation centre (ECIC) Eastman Dental Institute., London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobsen S, Petersen J, Ullman S, Junker P, Voss A, Rasmussen JM, Tarp U, Poulsen LH, van Overeem Hansen G, Skaarup B, Hansen TM, Podenphant J, Halberg P. A multicentre study of 513 Danish patients with systemic lupus erythematosus. II. Disease mortality and clinical factors of prognostic value. Clin Rheumatol. 1998;17(6):478-84. doi: 10.1007/BF01451283. PMID 9890675
- [Background] Bartels CM, Buhr KA, Goldberg JW, Bell CL, Visekruna M, Nekkanti S, Greenlee RT. Mortality and cardiovascular burden of systemic lupus erythematosus in a US population-based cohort. J Rheumatol. 2014 Apr;41(4):680-7. doi: 10.3899/jrheum.130874. Epub 2014 Feb 15. PMID 24532834
- [Background] Urowitz MB, Bookman AA, Koehler BE, Gordon DA, Smythe HA, Ogryzlo MA. The bimodal mortality pattern of systemic lupus erythematosus. Am J Med. 1976 Feb;60(2):221-5. doi: 10.1016/0002-9343(76)90431-9. PMID 1251849
- [Background] Cervera R, Khamashta MA, Font J, Sebastiani GD, Gil A, Lavilla P, Mejia JC, Aydintug AO, Chwalinska-Sadowska H, de Ramon E, Fernandez-Nebro A, Galeazzi M, Valen M, Mathieu A, Houssiau F, Caro N, Alba P, Ramos-Casals M, Ingelmo M, Hughes GR; European Working Party on Systemic Lupus Erythematosus. Morbidity and mortality in systemic lupus erythematosus during a 10-year period: a comparison of early and late manifestations in a cohort of 1,000 patients. Medicine (Baltimore). 2003 Sep;82(5):299-308. doi: 10.1097/01.md.0000091181.93122.55. PMID 14530779
- [Background] Doria A, Iaccarino L, Ghirardello A, Zampieri S, Arienti S, Sarzi-Puttini P, Atzeni F, Piccoli A, Todesco S. Long-term prognosis and causes of death in systemic lupus erythematosus. Am J Med. 2006 Aug;119(8):700-6. doi: 10.1016/j.amjmed.2005.11.034. PMID 16887417
- [Background] Manzi S, Meilahn EN, Rairie JE, Conte CG, Medsger TA Jr, Jansen-McWilliams L, D'Agostino RB, Kuller LH. Age-specific incidence rates of myocardial infarction and angina in women with systemic lupus erythematosus: comparison with the Framingham Study. Am J Epidemiol. 1997 Mar 1;145(5):408-15. doi: 10.1093/oxfordjournals.aje.a009122. PMID 9048514
- [Background] Skamra C, Ramsey-Goldman R. Management of cardiovascular complications in systemic lupus erythematosus. Int J Clin Rheumtol. 2010 Feb 1;5(1):75-100. doi: 10.2217/ijr.09.73. PMID 20305727
- [Background] Bruce IN, Gladman DD, Urowitz MB. Premature atherosclerosis in systemic lupus erythematosus. Rheum Dis Clin North Am. 2000 May;26(2):257-78. doi: 10.1016/s0889-857x(05)70138-1. PMID 10768212
- [Background] Salmon JE, Roman MJ. Accelerated atherosclerosis in systemic lupus erythematosus: implications for patient management. Curr Opin Rheumatol. 2001 Sep;13(5):341-4. doi: 10.1097/00002281-200109000-00001. PMID 11604586
- [Background] Asanuma Y, Oeser A, Shintani AK, Turner E, Olsen N, Fazio S, Linton MF, Raggi P, Stein CM. Premature coronary-artery atherosclerosis in systemic lupus erythematosus. N Engl J Med. 2003 Dec 18;349(25):2407-15. doi: 10.1056/NEJMoa035611. PMID 14681506
- [Background] Doria A, Shoenfeld Y, Wu R, Gambari PF, Puato M, Ghirardello A, Gilburd B, Corbanese S, Patnaik M, Zampieri S, Peter JB, Favaretto E, Iaccarino L, Sherer Y, Todesco S, Pauletto P. Risk factors for subclinical atherosclerosis in a prospective cohort of patients with systemic lupus erythematosus. Ann Rheum Dis. 2003 Nov;62(11):1071-7. doi: 10.1136/ard.62.11.1071. PMID 14583570
- [Background] Korkmaz H, Onalan O. Evaluation of endothelial dysfunction: flow-mediated dilation. Endothelium. 2008 Jul-Aug;15(4):157-63. doi: 10.1080/10623320802228872. PMID 18663619
- [Background] Inoue T, Node K. Vascular failure: A new clinical entity for vascular disease. J Hypertens. 2006 Nov;24(11):2121-30. doi: 10.1097/01.hjh.0000249684.76296.4f. PMID 17053528
- [Background] Halcox JP, Schenke WH, Zalos G, Mincemoyer R, Prasad A, Waclawiw MA, Nour KR, Quyyumi AA. Prognostic value of coronary vascular endothelial dysfunction. Circulation. 2002 Aug 6;106(6):653-8. doi: 10.1161/01.cir.0000025404.78001.d8. PMID 12163423
- [Background] Matsuzawa Y, Lerman A. Endothelial dysfunction and coronary artery disease: assessment, prognosis, and treatment. Coron Artery Dis. 2014 Dec;25(8):713-24. doi: 10.1097/MCA.0000000000000178. PMID 25365643
- [Background] Liao JK, Bettmann MA, Sandor T, Tucker JI, Coleman SM, Creager MA. Differential impairment of vasodilator responsiveness of peripheral resistance and conduit vessels in humans with atherosclerosis. Circ Res. 1991 Apr;68(4):1027-34. doi: 10.1161/01.res.68.4.1027. PMID 2009605
- [Background] Drexler H. Endothelial dysfunction: clinical implications. Prog Cardiovasc Dis. 1997 Jan-Feb;39(4):287-324. doi: 10.1016/s0033-0620(97)80030-8. PMID 9050817
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Piper MK, Raza K, Nuttall SL, Stevens R, Toescu V, Heaton S, Gardner-Medwin J, Hiller L, Martin U, Townend J, Bacon PA, Gordon C. Impaired endothelial function in systemic lupus erythematosus. Lupus. 2007;16(2):84-8. doi: 10.1177/0961203306074842. PMID 17402363
- [Background] Mak A, Kow NY, Schwarz H, Gong L, Tay SH, Ling LH. Endothelial dysfunction in systemic lupus erythematosus - a case-control study and an updated meta-analysis and meta-regression. Sci Rep. 2017 Aug 4;7(1):7320. doi: 10.1038/s41598-017-07574-1. PMID 28779080
- [Background] Libby P, Ridker PM, Hansson GK; Leducq Transatlantic Network on Atherothrombosis. Inflammation in atherosclerosis: from pathophysiology to practice. J Am Coll Cardiol. 2009 Dec 1;54(23):2129-38. doi: 10.1016/j.jacc.2009.09.009. PMID 19942084
- [Background] Petersen PE, Bourgeois D, Ogawa H, Estupinan-Day S, Ndiaye C. The global burden of oral diseases and risks to oral health. Bull World Health Organ. 2005 Sep;83(9):661-9. Epub 2005 Sep 30. PMID 16211157
- [Background] Albandar JM, Rams TE. Global epidemiology of periodontal diseases: an overview. Periodontol 2000. 2002;29:7-10. doi: 10.1034/j.1600-0757.2002.290101.x. No abstract available. PMID 12102700
- [Background] D'Aiuto F, Graziani F, Tete S, Gabriele M, Tonetti MS. Periodontitis: from local infection to systemic diseases. Int J Immunopathol Pharmacol. 2005 Jul-Sep;18(3 Suppl):1-11. PMID 16848982
- [Background] Noack B, Genco RJ, Trevisan M, Grossi S, Zambon JJ, De Nardin E. Periodontal infections contribute to elevated systemic C-reactive protein level. J Periodontol. 2001 Sep;72(9):1221-7. doi: 10.1902/jop.2000.72.9.1221. PMID 11577954
- [Background] D'Aiuto F, Orlandi M, Gunsolley JC. Evidence that periodontal treatment improves biomarkers and CVD outcomes. J Periodontol. 2013 Apr;84(4 Suppl):S85-S105. doi: 10.1902/jop.2013.134007. PMID 23631587
- [Background] Orlandi M, Suvan J, Petrie A, Donos N, Masi S, Hingorani A, Deanfield J, D'Aiuto F. Association between periodontal disease and its treatment, flow-mediated dilatation and carotid intima-media thickness: a systematic review and meta-analysis. Atherosclerosis. 2014 Sep;236(1):39-46. doi: 10.1016/j.atherosclerosis.2014.06.002. Epub 2014 Jun 17. PMID 25014033
- [Background] D'Aiuto F, Nibali L, Parkar M, Patel K, Suvan J, Donos N. Oxidative stress, systemic inflammation, and severe periodontitis. J Dent Res. 2010 Nov;89(11):1241-6. doi: 10.1177/0022034510375830. Epub 2010 Aug 25. PMID 20739696
- [Background] Tonetti MS, D'Aiuto F, Nibali L, Donald A, Storry C, Parkar M, Suvan J, Hingorani AD, Vallance P, Deanfield J. Treatment of periodontitis and endothelial function. N Engl J Med. 2007 Mar 1;356(9):911-20. doi: 10.1056/NEJMoa063186. PMID 17329698
- [Background] de Pablo P, Dietrich T, McAlindon TE. Association of periodontal disease and tooth loss with rheumatoid arthritis in the US population. J Rheumatol. 2008 Jan;35(1):70-6. Epub 2007 Nov 15. PMID 18050377
- [Background] Calderaro DC, Ferreira GA, de Mendonca SM, Correa JD, Santos FX, Sancao JG, da Silva TA, Teixeira AL. Is there an association between systemic lupus erythematosus and periodontal disease? Rev Bras Reumatol Engl Ed. 2016 May-Jun;56(3):280-4. doi: 10.1016/j.rbre.2015.08.003. Epub 2015 Sep 8. English, Portuguese. PMID 27267648
- [Background] Rutter-Locher Z, Smith TO, Giles I, Sofat N. Association between Systemic Lupus Erythematosus and Periodontitis: A Systematic Review and Meta-analysis. Front Immunol. 2017 Oct 17;8:1295. doi: 10.3389/fimmu.2017.01295. eCollection 2017. PMID 29089946
- [Background] Ryden L, Buhlin K, Ekstrand E, de Faire U, Gustafsson A, Holmer J, Kjellstrom B, Lindahl B, Norhammar A, Nygren A, Nasman P, Rathnayake N, Svenungsson E, Klinge B. Periodontitis Increases the Risk of a First Myocardial Infarction: A Report From the PAROKRANK Study. Circulation. 2016 Feb 9;133(6):576-83. doi: 10.1161/CIRCULATIONAHA.115.020324. Epub 2016 Jan 13. PMID 26762521
- [Background] Fabbri C, Fuller R, Bonfa E, Guedes LK, D'Alleva PS, Borba EF. Periodontitis treatment improves systemic lupus erythematosus response to immunosuppressive therapy. Clin Rheumatol. 2014 Apr;33(4):505-9. doi: 10.1007/s10067-013-2473-2. Epub 2014 Jan 11. PMID 24415114